CLINICAL TRIAL: NCT01748656
Title: Comparison of Two Noninvasive Positive Pressure Ventilation Devices Using Target Volume Modes in Obesity Hypoventilation Syndrome (OHS): A Pilot Randomized Crossover Controlled Trial
Brief Title: Target Volume in Noninvasive Positive Pressure Ventilation
Acronym: CIBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-AGIR-02
Record Dates: First submitted 2012-12-11; First posted 2012-12-12 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2012-12

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: Noninvasive ventilation; Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVAPS (Active Comparator): AVAPS mode(BIPAP-A30-PHILIPS-RESPIRONICS)1 night
  Interventions: Device: IVAPS
- IVAPS (Active Comparator): IVAPS mode(STELAR 150-RESMED)1 night
  Interventions: Device: AVAPS

INTERVENTIONS:
Device: IVAPS — IVAPS mode (RESMED Stelar 150) during 1 night
  Arms: AVAPS
Device: AVAPS — AVAPS mode (PHILIPS-RESPIRONICS-A30) during 1 night
  Arms: IVAPS

SUMMARY:
Patients with OHS are efficiently managed with long term home-based nocturnal noninvasive positive pressure ventilation (NIPPV). Several NIPPV devices offer the feature of automatically adjusting pressure support (and/or respiratory back-up rate) on the basis of a pre-determined "ideal tidal volume" or "ideal ventilation". However algorithms used to achieve these ideal targets are different among different commercialized devices and the relative efficacy from an algorithm compared to another remains unknown. The main objective is this study is to compare two commercialized NIPPV that have this option

DETAILED DESCRIPTION:
RESMED Stellar-150 (IVAPS mode)versus PHILIPS-RESPIRONICS A30 (AVAPS-mode).

ELIGIBILITY:
Inclusion Criteria:

* Patient with Obesity hypoventilation Syndrome (BMI≥ 30 kg/m2 and diurnal PaCO2 ≥ 45mmHg at diagnosis after exclusion of others causes of hypoventilation)
* 18 to 75 years old
* In stable state but treated by nocturnal NIPPV for more than 3 months and adherent to NIPPV (above 4h/night).

Exclusion Criteria:

* patient treated with additional long term Oxygen therapy
* Patient previously treated by AVAPS mode or IVAPS mode

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Mean Nocturnal transcutaneous CO2 pressure (Mean nocturnal PtCO2) | 1 night
  transcutaneous CO2 pressure is measured overnight. It is a reliable estimation of arterial PaCO2 to monitor nocturnal ventilation in adults with chronic respiratory failure.

SECONDARY OUTCOMES:
Mean transcutaneous CO2 pressure during REM Sleep | 1 Night
Mean nocturnal SpO2 | 1 night
Awake arterial PaCO2 after 1 hour of NIPPV withdrawal | After 1 night
Micro-arousals/hour of sleep | 1 night
Sleep Quality assess by Visual analogic scale (100mm) | 1 night
Respiratory residual events detected by NIPPV built-in softwares | 1 Night

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pepin, MD PHD, Principal Investigator — CHU Grenoble France
Locations (1):
- Sleep Laboratory, Grenoble Univeristy Hospital, Grenoble, France